CLINICAL TRIAL: NCT00208858
Title: Nicotine Craving: Neural Correlates of Treatment Effect - A Pilot Study
Brief Title: A Pilot Study of the Neural Correlates of Treatment Effect on Nicotine Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Karen Drexler, Asc Professor/Director, Substance Abuse Treatment, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0624-2004; DA00366-02 (Other: Other); TPN-100 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to gather pilot data to determine feasibility of and guide the development of a larger clinical trial investigating the effects of topiramate as an adjunct to nicotine replacement therapy and behavioral counseling in smoking cessation treatment. It is hypothesized that topiramate will decrease nicotine craving and result in improved outcomes for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Male, between ages of 18-55
* Meets DSM-IV criteria for nicotine dependence
* Smoke at least 20 cigarettes per day
* Motivated to quit smoking

Exclusion Criteria:

* Serious or unstable medical conditions
* Current psychiatric disorder requiring medication or treatment
* Taking medication that create risk of interaction with study drug
* Current participation in another smoking cessation treatment

Ages: 18 Years to 55 Years | Sex: Male
Age Groups: Adult
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Drexler, MD, Principal Investigator — Emory University, Atlanta VA Medical Center
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States